CLINICAL TRIAL: NCT04690790
Title: Pulmonary Nodule Localization Under Thoracoscopic Surgery- a Machine Learning Based Retrospective Analysis and Prospective Validation
Brief Title: Pulmonary Nodule Localization Prospective Validation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Tu, Yuan-Kun, president, E-DA Hospital
Other Study IDs: EMRP56109N
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Video-assisted Thoracic Surgery; Pulmonary Nodules
Keywords: Video-assisted thoracic surgery; Thoracoscopy; Localization; Pulmonary nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules | interventions — Thoracoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracoscopy — Patients who are indicated for thoracoscopic nodulectomy.

SUMMARY:
Localization is the key for successful excision of small target nodules under thoracoscopy, but the procedure also brings risks to patients. However, the criteria is still unclear. The investigators will validate the prediction model produced by institutional retrospective analysis in the prospective cohort.

DETAILED DESCRIPTION:
Excision of targeted lung nodules during thoracoscopy sometimes needs placing a mark before surgery. The procedure of mark placement (localization) could probably cause damages to the patients. However, the criteria for patient selection is still not clear. Through respective analysis, the investigators have set up a prediction model and wish to validate this model prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20 years
* Lung nodule size ≦2cm on the pre-operative computed tomography (CT)
* Nodulectomy is performed under thoracoscopy

Exclusion Criteria:

* Age < 20 years
* Lung nodule size > 2cm on CT or in the final pathology report
* Open surgery for nodulectomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for thoracoscopic nodulectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Nodule detection | During surgery
  Whether the nodule could be detected by conventional visualization or palpation

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Wei Kao, M.D., M.S., Principal Investigator — E-DA Hospital
Locations (1):
- E-DA Hospital, Kaohsiung City, Taiwan